CLINICAL TRIAL: NCT03438734
Title: Comparison of Low Versus Normal Flow Anesthesia on Cerebral Oxygenation and Bispectral Index in Morbidly Obese Patients Undergoing Sleeve Gastrectomy: Prospective, Randomized Clinical Trial
Brief Title: Comparison of Low Versus Normal Flow Anesthesia on Cerebral Oxygenation and Bispectral Index in Morbidly Obese Patients
Acronym: CerOxygen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sedat AKBAS, Asst. Prof., Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: sedatakbas1
Record Dates: First submitted 2018-02-06; First posted 2018-02-20 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Morbid Obesity; Anesthesia Awareness; Anesthesia Complication
Keywords: Bariatric surgery; Low flow anesthesia; Bispectral index; Regional cerebral oximetry
MeSH Terms: conditions — Obesity, Morbid; Intraoperative Awareness | interventions — Spectroscopy, Near-Infrared; Consciousness Monitors

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical Study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low flow (Active Comparator): Anesthesia was maintained with desflurane inhalation with a flow of 2 L/min in 0.5 O2 oxygen-air mixture in both groups. While target minimum alveolar concentration (MAC) was 1-1.5 and the flow rate was adjusted to 0.75 L/min. Regional cerebral oxygen saturation is a useful clinical research tool for noninvasive and continuous monitoring of hemodynamic and brain oxygenation. Regional cerebral oxygen saturation (Near-infrared spectroscopy system, NIRS, Cerebral Oximeter) monitoring was performed to all patients.
  The most effective method for depth of anesthesia and assessment of sedation is bispectral analysis of mean frequency of electroencephalography. The values of Bispectral Index (BIS, Bispectral Index, Monitoring System) decreases with the deepening of anesthesia.
  Interventions: Device: Regional cerebral oxygen saturation; Device: Bispectral Index (BIS)
- Normal flow (Sham Comparator): Anesthesia was maintained with desflurane inhalation with a flow of 2 L/min in 0.5 O2 oxygen-air mixture in both groups. While target minimum alveolar concentration (MAC) was 1-1.5 and the flow rate was adjusted to 1.5 L/min.Regional cerebral oxygen saturation is a useful clinical research tool for noninvasive and continuous monitoring of hemodynamic and brain oxygenation. Regional cerebral oxygen saturation (Near-infrared spectroscopy system, NIRS, Cerebral Oximeter) monitoring was performed to all patients.
  The most effective method for depth of anesthesia and assessment of sedation is bispectral analysis of mean frequency of electroencephalography. The values of Bispectral Index (BIS, Bispectral Index, Monitoring System) decreases with the deepening of anesthesia.
  Interventions: Device: Regional cerebral oxygen saturation; Device: Bispectral Index (BIS)

INTERVENTIONS:
Device: Regional cerebral oxygen saturation — Regional cerebral oxygen saturation is a useful clinical research tool for noninvasive and continuous monitoring of hemodynamic and brain oxygenation. Regional cerebral oxygen saturation (Near-infrared spectroscopy system, NIRS, Cerebral Oximeter) monitoring was performed to all patients.
  Other Names: NIRS (Near-infrared spectroscopy system)
Device: Bispectral Index (BIS) — The most effective method for depth of anesthesia and assessment of sedation is bispectral analysis of mean frequency of electroencephalography. The values of BIS decreases with the deepening of anesthesia.
  Other Names: BIS

SUMMARY:
Obesity is a chronic disease that affects quality and duration of life negatively. It's not clearly known the effects of low flow anesthesia on cerebral oxygenation with high-risk morbidly obese patients. In this study, it was aimed to compare the effects of general anesthesia with low flow (0,75 L/min) and normal flow (1,5 L/min) on cerebral oxygenation and depth of anesthesia in morbidly obese patients in bariatric surgery.

DETAILED DESCRIPTION:
Obesity is a chronic disease that affects quality and duration of life negatively. It is one of the most important health problem in the world along with very common in Turkey. Initially, obesity was considered the problem of developed countries but it has become inevitable with increase income levels, changes in lifestyles, reduction of energy consumption and increase of energy intake in developing countries. Today, the second important cause of preventable deaths after smoking is obesity. The World Health Organization (WHO) has stated that it will be the most important health problem of the 21st century. According to WHO determinations; as of 2008, the prevalence of overweight in the world is 35% and the prevalence of obesity is around 11%. The definition of body mass index (BMI) is used in defining and classifying obesity. WHO is making the definition of overweight and obesity based on body mass index [BMI = Weight (kg) / Height (m2)]. It is called as obesity when the calculated value is over 30 kg/m2, morbid obesity over 40 kg/m2 and super obesity over 50 kg/m2.

Morbid obesity operations, with effective results on achieving weight loss continuity once it has been widely applied in Europe and the United States, have been frequently implemented in Turkey as well. With the rising obesity in Turkey, laparoscopic bariatric surgery which has low complication rates is preferred.

Low flow general anesthesia is applied to reduce pollution rates and treatment costs in operation rooms. However, the reduction of fresh gas flow should not affect the quality and safety of anesthesia management, especially in high risk operations such as morbid obesity surgery. Insufflation of abdominal cavity with carbon dioxide during laparoscopic surgery is resulted in increased intraabdominal pressure, decreased functional residual capacity and pulmonary compliance, increased hypercapnia and systemic vascular resistance. Especially in the trendelenburg position it may be difficult to detect cerebral hypoxia as a consequence of increased intracranial pressure and decreased cerebral blood flow .

During general anesthesia, there are several options for monitoring the cerebral condition. One of them is cerebral oximetry method which estimates regional tissue oxygenation by transcutaneous measurement on the frontal cortex. Near-infrared spectroscopy (NIRS) is a monitor used following the adequacy of cerebral perfusion with noninvasive and continuous measurement and reflects regional saturation.

With the development of technology, the safety of anesthesia devices and the advancement of monitoring techniques are positively affecting the anesthesia management. The effects of low flow anesthesia, which has been used for years and whose positive aspects are well practiced, are not clearly known on cerebral oxygenation with high-risk morbidly obese patients. In this prospective randomized study, it was aimed to compare the effects of general anesthesia with low flow (0,75 L/min) and normal flow (1,5 L/min) on cerebral oxygenation and depth of anesthesia in morbidly obese patients in bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology score I-III,
* 18-65 years,
* BMI> 35

Exclusion Criteria:

* American Society of Anesthesiology IV,
* Under 18 years,
* Over 65 years,
* Obstetric patients,
* Uncontrolled diabetes mellitus, cardiovascular and pulmonary disease,
* Cerebrovascular disease,
* Patients who refused informed consent forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65 years
Enrollment: 52 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-02-17 (Actual)

PRIMARY OUTCOMES:
Regional Cerebral Oxygen Saturations (Left and Right) | From beginning of anesthesia (15 minutes before anesthesia) to end of anesthesia (15 minutes after anesthesia) up to nearly 5 hours
  The measurement of Regional Cerebral Oxygen Saturations by cerebral oximetry method which estimates regional tissue oxygenation by transcutaneous measurement on the frontal cortex. Cerebral oximeter (or named as NIRS, Near-infrared spectroscopy) is a monitor used following the adequacy of cerebral perfusion with noninvasive and continuous measurement and reflects regional saturation

SECONDARY OUTCOMES:
Heart rate | From beginning of anesthesia (15 minutes before anesthesia) to end of anesthesia (15 minutes after anesthesia) up to nearly 5 hours
  Heart rate (beat/min)
Systolic and Diastolic Arterial Pressure (both) | From beginning of anesthesia (15 minutes before anesthesia) to end of anesthesia (15 minutes after anesthesia) up to nearly 5 hours
  Systolic and Diastolic Arterial Pressure (both) (mmHg)
End-tidal carbon dioxide (EtCO2) | From beginning of anesthesia (15 minutes before anesthesia) to end of anesthesia (15 minutes after anesthesia) up to nearly 5 hours
  EtCO2 is the measurement of the exhaled CO2 by capnography. This value is expressed in millimeters of mercury (mmHg) of CO2.
Bispectral Index (BIS) | From beginning of anesthesia (15 minutes before anesthesia) to end of anesthesia (15 minutes after anesthesia) up to nearly 5 hours
  Bispectral Index is a method for depth of anesthesia and assessment of sedation. The values of BIS decreases with the deepening of anesthesia. The values of 40-60 characterize the appropriate depth of anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Sedat AKBAS, Study Director — Inonu University Medical Faculty
Locations (1):
- Sedat AKBAS, Malatya, Türkiye-Türkçe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones KB Jr. Experience with the Roux-en-Y gastric bypass, and commentary on current trends. Obes Surg. 2000 Apr;10(2):183-5. doi: 10.1381/096089200321668659. No abstract available. PMID 10782184
- [Background] Vegh T. Cerebral Oximetry in General Anaesthesia. Turk J Anaesthesiol Reanim. 2016 Oct;44(5):247-249. doi: 10.5152/TJAR.2016.26092016. Epub 2016 Oct 1. No abstract available. PMID 27909605
- [Result] Kupisiak J, Goch R, Polenceusz W, Szyca R, Leksowski K. Bispectral index and cerebral oximetry in low-flow and high-flow rate anaesthesia during laparoscopic cholecystectomy - a randomized controlled trial. Wideochir Inne Tech Maloinwazyjne. 2011 Dec;6(4):226-30. doi: 10.5114/wiitm.2011.26256. Epub 2011 Dec 20. PMID 23255984

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT03438734/Prot_SAP_000.pdf